CLINICAL TRIAL: NCT00279097
Title: A Safety Study to Evaluate Intracranial Pressure With the Utilization of High Frequency Chest Wall Oscillation (HFCWO) Using the Vest™ on Mechanically Ventilated Neurosurgical Patients
Brief Title: Safety Study to Evaluate Intracranial Pressure During High Frequency Chest Wall Oscillation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Hill-Rom (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR-0038
Record Dates: First submitted 2006-01-17; First posted 2006-01-19 (Estimated); Last update posted 2006-11-16 (Estimated); Status verified 2006-11

CONDITIONS: Intracranial Pressure
Keywords: Intracranial pressure; High Frequency Chest Wall Oscillation; Neurosurgery
MeSH Terms: interventions — Chest Wall Oscillation

INTERVENTIONS:
Device: High Frequency Chest Wall Oscillation

SUMMARY:
The purpose of this study is to evaluate changes in intracranial pressure (ICP) during or immediately following high frequency chest wall oscillation (HFCWO) treatment with the Vest™ in neurosurgical subjects.

DETAILED DESCRIPTION:
This study is a single site safety study to evaluate changes in intracranial pressure during or immediately following HFCWO treatment with the Vest™ in neurosurgical subjects with intracranial pressure monitors having normal opening pressures and ICP less than or equal to 20 mmHg. The secondary objective of this study is to evaluate changes in arterial blood gases that may result with Vest™ therapy in ventilated patients.

ELIGIBILITY:
Inclusion Criteria:

* ICP monitor with normal opening pressure (greater than or equal to 20 mmHg)
* On ventilator
* Arterial line in place
* Age equal to or greater than 18
* Admitted to neurotrauma intensive care unit (ICU)

Exclusion Criteria:

* Inability to obtain informed consent
* Unstable spinal cord injury
* ICP > 20 mmHg sustained for > 5 minutes
* Hemodynamic instability within the prior 12 hours
* Active hemoptysis
* Hemothorax
* New onset, unstable arrhythmia
* Enrollment in another interventional study
* Aneurysm that has not been clipped or coiled
* Coagulopathic head injury subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2006-01; Study Completion 2006-09

PRIMARY OUTCOMES:
Intracranial pressure
SpO2
Heart rate
Mean arterial pressure (MAP)
Arterial blood gases (ABGs)

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Levine, MD, Principal Investigator — University of Texas
Locations (1):
- University of Texas at Houston/Memorial Hermann Hospital, Houston, Texas, United States